CLINICAL TRIAL: NCT00004146
Title: Phase II Clinical and Pharmacologic Study of Radiation Therapy and CAI (Carboxy-Amido Triazole) in Adults With Newly Diagnosed Glioblastoma Multiforme
Brief Title: Carboxyamidotriazole + RT in Treating Patients Newly Diagnosed Supratentorial GBM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-03011; NCI-2012-03011 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR67378; NABTT-9904 (Other: New Approaches to Brain Tumor Therapy Consortium); NABTT-9904 (Other: CTEP); U01CA062475 (NIH)
Record Dates: First submitted 1999-12-10; First posted 2004-06-04 (Estimated); Results first posted 2015-05-08 (Estimated); Last update posted 2015-05-08 (Estimated); Status verified 2015-04

CONDITIONS: Adult Giant Cell Glioblastoma; Adult Glioblastoma; Adult Gliosarcoma
MeSH Terms: conditions — Glioblastoma; Gliosarcoma | interventions — Radiotherapy; Radiation; carboxyamido-triazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (RT and CAI) (Experimental): Patients receive induction therapy consisting of radiotherapy once daily 5 days a week plus oral carboxyamidotriazole once daily for 6 weeks followed by carboxyamidotriazole alone daily for 4 weeks. Patients continue on oral carboxyamidotriazole once daily as maintenance therapy in the absence of disease progression or unacceptable toxicity. Patients are followed monthly for survival.
  Other: pharmacological study, radiation therapy
  Interventions: Radiation: radiation therapy; Drug: carboxyamidotriazole; Other: pharmacological study

INTERVENTIONS:
Radiation: radiation therapy — Undergo radiotherapy
  Other Names: irradiation; radiotherapy; therapy, radiation
Drug: carboxyamidotriazole — Given orally
  Other Names: CAI; carboxyamido-triazole; carboxyaminoimidazole
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Combining radiation therapy with chemotherapy may kill more tumor cells. Phase II trial to study the effectiveness of carboxyamidotriazole plus radiation therapy in treating patients who have newly diagnosed supratentorial glioblastoma multiforme.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate overall survival rate in patients administered CAI (carboxyamidotriazole) and radiation therapy to adults with newly diagnosed glioblastoma multiforme.

II. To determine the toxicity of CAI when combined with cranial irradiation. III. To estimate correlations between pharmacokinetic parameters, including steady state CAI concentration, with toxicity and/or drug activity in this patient population.

IV. To estimate duration of disease free progression with this treatment regime.

OUTLINE: This is a multicenter study.

Patients receive induction therapy consisting of radiotherapy once daily 5 days a week plus oral carboxyamidotriazole once daily for 6 weeks followed by carboxyamidotriazole alone daily for 4 weeks. Patients continue on oral carboxyamidotriazole once daily as maintenance therapy in the absence of disease progression or unacceptable toxicity. Patients are followed monthly for survival.

PROJECTED ACCRUAL: A total of 54 patients will be accrued for this study over 1.5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed supratentorial grade IV astrocytoma (glioblastoma multiforme)
* Patients must have measurable or non-measurable tumor on the post operative, pretreatment MRI/CT scan (within two weeks of starting treatment)
* Patients must not have received prior radiation therapy, chemotherapy, hormonal therapy, immunotherapy or therapy with biologic agents (including immunotoxins, immunoconjugates, antisense, peptide receptor antagonists, interferons, interleukins, TIL, LAK or gene therapy), or hormonal therapy for their brain tumor; glucocorticoid therapy is allowed
* Patients must have recovered from the immediate post-operative period and be maintained on a stable steroid regimen (no increase for the last five days)
* Absolute neutrophil count >= 1500/mm^3
* Platelets >= 100,000/mm^3
* Hemoglobin concentration >= 9.0 g/dl
* Creatinine =< 1.7mg/dL
* Total bilirubin =< 1.2 mg/dl
* Transaminases =< 2 times above the upper limits of the institutional normal
* Estimated life expectancy greater than 2 months
* Patients must give informed consent and understand the investigational nature of this study and its potential risks and benefits
* Patients, if female and of childbearing potential must have a negative serum beta-hCG test and must not be breast feeding; all patients with the potential for pregnancy should be counseled and requested to follow acceptable birth control methods to avoid conception
* Patients must have a Karnofsky performance status of >= 60%
* No other serious concurrent infection or other medical illness should be present which would jeopardize the ability of the patient to receive the drug outlined in this protocol with reasonable safety
* Patients must have no concurrent malignancy except curatively treated basal or squamous cell carcinoma of the skin or carcinoma in situ; patients with prior malignancies must be disease-free for >= five years

Exclusion Criteria:

* Patients must be able to comply with prescribed medical care
* Prior therapy for the brain tumor (except surgery)
* Prior treatment with antineoplastic agents, including CAI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2000-03; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tom Mikkelsen, MD, Principal Investigator — New Approaches to Brain Tumor Therapy Consortium
Locations (8):
- United States (8):
  - University of Alabama Birmingham, Birmingham, Alabama
  - Moffitt Cancer Center, Tampa, Florida
  - Emory University/Winship Cancer Institute, Atlanta, Georgia
  - Johns Hopkins University, Baltimore, Maryland
  - Henry Ford Hospital, Detroit, Michigan
  - Wake Forest University, Winston-Salem, North Carolina
  - University of Pennsylavania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between March and October of 2000 55 patients(pts) were accrued from outpatient clinics throughout ABTC(Adult Brain Tumor Consortium) consortium clinics
Pre-assignment Details: pts had to have confirmed GBM (Glioblastoma) and be untreated except for biopsy or surgery and corticosteroids.
Groups:
- CAI With RT - Arm 1: CAI with RT
  carboxyamidotriazole :
  CAI : CAI 250 mg PO plus RT followed by 4wks CAI alone followed by 8wks CAI then MRI if stable or better continue until progression and then follow for survival
  radiation therapy :
Period: Overall Study
Arm/Group | CAI With RT - Arm 1
Started | 55
Completed | 55
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | CAI With RT - Arm 1
Number analyzed (Participants) | 55
Age, Customized [Median (Full Range); unit: years] | 59 [31.0 to 79.4]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 33
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 54
  More than one race | 0
  Unknown or Not Reported | 0
Karnofsky Performance Status [Number; unit: participants] — performance status is an attempt to quantify patients' general well-being and activities of daily life. The scale is in intervals of 10. 100 being normal and 0 dead. For ABTC studies you had to have a KPS of at least 60 (Requires occasional assistance, but is able to care for most of his personal needs) to be eligible for the study.
  participants
    Performance Status 100 | 9
    Performance Status 90 | 24
    Performance Status 80 | 10
    Performance Status 70 | 10
    Performance Status 60 | 2

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival Rate
Description: estimated period of time event assessed 30 months. event assessed from time of histological diagnosis to death
Time Frame: approximately 30 months
Population: intent to treat pt population. time from histological diagnosis to death.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | CAI With RT - Arm 1
Number analyzed (Participants) | 55
months | 10.3 [8.5 to 12.8]
Statistical Analysis 1: Comparison: CAI With RT - Arm 1; the study design is to detect 30% reduction in hazard of deaths with 78% power at one side alpha level of 0.10. Overall survial time was calculated from time of histological diagnosis until time of death from any event; Test type: Superiority or Other; p = 0.10, t-test, 1 sided; Hazard Ratio (HR) = 0.85, 95% CI 2-sided [0.65 to 1.12]

2. Primary Outcome: Toxicity of CAI When Combined With RT
Description: patients who experienced a grade 3 or higher event considered at least possibly related to CAI
Time Frame: pts were reviewed for toxicity while on treatement - median time of 2 months
Population: pts were treated for a median time of 2 months (23 days to 46 months). patients who experienced a grade 3 or higher event considered at least possibly related to CAI
Measure: Number; unit: participants
Arm/Group | CAI With RT - Arm 1
Number analyzed (Participants) | 55
participants | 16

3. Primary Outcome: Correlation Between PK CAI and Toxicity in This pt Population
Description: PK paramenters including steady state CAI concentrations with toxicity/or drug activity
Time Frame: during treatment
Population: 50 subjects had PK samples for analysis
Measure: Mean (Standard Deviation); unit: ug/ml
Groups:
- CAI With RT + Enzyme Inducing Anticonvulsants; CAI With RT Without Enzyme Inducing Anticonvulsants: CAI with RT
  carboxyamidotriazole :
  CAI : CAI 250 mg PO plus RT followed by 4wks CAI alone followed by 8wks CAI then MRI if stable or better continue until progression and then follow for survival
  radiation therapy :
Arm/Group | CAI With RT + Enzyme Inducing Anticonvulsants | CAI With RT Without Enzyme Inducing Anticonvulsants
Number analyzed (Participants) | 42 | 8
ug/ml | 1.3 (1.22) | 4.06 (1.5)

ADVERSE EVENTS:
Time Frame: AE were collected while patients were on active treatment and for 30 days following treatment. pts were on active treatment for a median time of 2 months (23 days - 46 months)
Groups:
- Arm 1: CAI with RT
  carboxyamidotriazole :
  CAI : CAI 250 mg PO plus RT followed by 4wks CAI alone followed by 8wks CAI then MRI if stable or better continue until progression and then follow for survival
  radiation therapy :
Arm/Group | Arm 1
Serious Adverse Events (participants affected / at risk) | 7/55
Other Adverse Events (participants affected / at risk) | 9/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=55)
aspartate aminotransferase (Investigations) | 1 (1)
Alanine aminotransferase (Investigations) | 1 (1)
febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
reversible vision loss (Eye disorders) | 2 (2)
hemorrhage-other (Gastrointestinal disorders) | 1 (1)
hyperuricemia (Metabolism and nutrition disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=55)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
fatigue (General disorders) | 5 (5)
anemia (Blood and lymphatic system disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less